CLINICAL TRIAL: NCT04253704
Title: Placebo-controlled Double-blinded Trial to Evaluate the Effects of Short-term (1-2 Weeks) Treatment With 2% (Isosorbide di-(Linoleate/Oleate)) (IDL) Lotion on Skin Hydration and Transepidermal Water Loss in Females With Dry Skin
Brief Title: Effects of 2% IDL Lotion on Skin Hydration and Transepidermal Water Loss in Females With Dry Skin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shyla Cantor (Industry)
Collaborators: Sytheon Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Shyla Cantor, Principal Investigator, Sytheon Ltd.
Organization: Sytheon Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYT.P0104-B1.B2
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Xerosis Cutis
Keywords: transepidermal water loss; skin hydration; vapometer; novameter

STUDY DESIGN:
Intervention Model Description: Test materials were applied to forearm skin of each subject. The left arm was used for the test material IDL lotion. The right arm was used for the hydrating control lotion.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants were not told which arm received treatment versus placebo lotions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 2% IDL lotion (Experimental): The left arm of each subject was used for the test material hydrating lotion (IDL).
  Interventions: Combination Product: IDL lotion
- Control lotion (Placebo Comparator): The right arm of each subject was used for control lotion lacking the IDL component.
  Interventions: Combination Product: Control lotion

INTERVENTIONS:
Combination Product: IDL lotion — IDL lotion is water-based (> 80%) with isosorbide di-(linoleate/oleate) (2.0%), caprylic/capric triglycerides (5%), glycerin (3%), glyceryl stearate (2.5%), dimethicone (2.0%), steareth-20 (1.5%), cetyl alcohol (1.0%), and butyrospermum parkii (shea) butter (1.0%).
  Other Names: IDL RC-02-38 / P0104-B1
  Arms: 2% IDL lotion
Combination Product: Control lotion — Control lotion is water-based (> 80%) with caprylic/capric triglycerides (5%), glycerin (3%), glyceryl stearate (2.5%), dimethicone (2.0%), steareth-20 (1.5%), cetyl alcohol (1.0%), and butyrospermum parkii (shea) butter (1.0%).
  Other Names: RC-02-38A / P0104-B2
  Arms: Control lotion

SUMMARY:
This was a placebo-controlled double-blinded trial to compare effects of 2% IDL lotion to placebo in female subjects with dry skin. Primary endpoints were skin hydration (NovaMeter) and transepidermal water loss (VapoMeter).

DETAILED DESCRIPTION:
1. Objective: To evaluate the efficacy of two topically applied test materials and the ability to increase hydration and decrease the transepidermal water loss of the skin. Efficacy was evaluated instrumentally using the NovaMeter and VapoMeter.
2. Test Material Description: On January 4, 2017, two test samples labeled Hydrating Lotion HydraSynol IDL RC-02-38, 12/21/16 and Hydrating Lotion Control RC-02-38A, 12/21/16 were received from Sytheon Ltd. and assigned CR Lab Nos.: P0104-B1 and P0104-B2, respectively.
3. Test Material Handling: Upon arrival at Cantor Research Laboratories, Inc., the test materials were assigned a unique laboratory code number and entered into a daily log identifying the lot number, sample description, sponsor, date received and tests requested. Samples are retained for a period of three months beyond submission of final report unless otherwise specified by the sponsor or if sample is known to be in support of governmental applications, in which case retained samples are kept two years beyond final report submission. Sample disposal is conducted in compliance with appropriate federal, state and local ordinances.
4. Recruitment: Panel selection was accomplished by advertisements in local periodicals, community bulletin boards, phone solicitation, electronic media or any combination thereof.
5. Informed Consent: In compliance with 21 CFR Ch.1 Part 50, Subpart B, informed consent was obtained from each volunteer prior to the commencement of the study. The consent form described the procedures, possible adverse effects, associated risks, and potential benefits of the study and the limits of liability. Panelists signed and dated the informed consent document to indicate their authorization to proceed and acknowledge their understanding of the contents.
6. NovaMeter: The Novameter is a multifunctional electronic laboratory instrument that measures skin impedance. It is designed to provide non-invasive, objective, reproducible method of measurement to quantify biophysical characteristics and relative hydration of the skin.
7. VapoMeter: The VapoMeter is a fully portable instrument for measureing TEWL (transepidermal water loss) values and evaporation rates. TEWL is an indicator of the skin's barrier function. The core of the VapoMeter is a sensitive humidity sensor that is inside a cylindrical measurement chamber. This chamber is closed by the skin or other measurement surface during the measurement period and is unaffected by ambient airflows. The sensor monitors the increase of relative humidity (RH) inside the chamber during the measurement. The evaporation rate value (g/m²h) is automatically calculated from the RH increase. The chamber is passively ventilated between measurements and the ventilation time is automatically controlled. The VapoMeter is widely accepted and an efficient instrument for TEWL measurements.
8. Washout period: Five days prior to the study the panelists were told to not use any moisturizers or treatment products on their arms and refrain from using any other products during the course of the study. They were asked to wash their arms with only ivory soap and pat dry.
9. Baseline: The panelists arrived at the lab with their arms washed by water alone (if forearm skin was not dry, the panelist was asked to wash their arms with only ivory soap and pat dry). Panelists with Skin Dryness Grade of 6 and 7 were inducted in the study. A trained technician examined the test areas (left and right volar arms) for any abnormalities that would obstruct the measurements. The left arm was used for the test material Hydrating Lotion HydraSynol IDL RC-02-38, 12/21/16 (CR Lab No. P0104-B1). The right arm was used for Hydrating Lotion Control RC-02-38A, 12/21/16 (CR Lab No. P0104-B2). The panelists were required to equilibrate to the controlled environment with a constant temperature of 70 degrees F and humidity of 30% Rh for half hour. Measurements on each arm (left and right volar arms) were taken using the NovaMeter and VapoMeter. A trained technician then applied each test material to the respective volar arm in order for the panelist to observe the manner in which the products should be applied for two weeks. The test materials were allowed to dry before the dismissal of the panelist. The panelists were then given the pre weighed test materials as well as a study diary in order to list the time of each application, the date and any subjective comments that they might have about the test materials.
10. Week 2: The panelists arrived at the lab with their arms applied with the test materials at least five hours prior. A trained technician examined the test areas (left and right volar arms) for any abnormalities that would obstruct the measurements. The panelists were allowed to equilibrate to the controlled environment with a constant temperature of 70 degrees F and humidity of 30% Rh for a half hour. Measurements on each arm (left and right volar arms) were taken again using the NovaMeter and VapoMeter. The test materials were weighed and diaries collected to check for compliance.
11. Day 18 (after 4 days regression): The panelists arrived at the lab. A trained technician examined the test areas (left and right volar arms) for any abnormalities that would obstruct the measurements. The panelists were allowed to equilibrate to the controlled environment with a constant temperature of 70 degrees F and humidity of 30% Rh for a half hour. Measurements on each arm (left and right volar arms) were taken again using the NovaMeter and VapoMeter.
12. Adverse reactions: Subjects were instructed to report any delayed reactions which might occur after the final reading. Clients are notified immediately in the case of an adverse reaction and a determination is made as to a treatment program if necessary.
13. Statistical Analysis: All of the data was tabulated in a Microsoft® Excel spreadsheet. Using the t-Test, the statistical significance of the net change from baseline (pre-application) to each subsequent time point was assessed. Statistical significance was defined at the p=0.05 or less level (corresponding to a 95% or greater confidence level).

ELIGIBILITY:
Inclusion Criteria:

1. Females who were thirty-five to fifty-seven years of age.
2. Individuals free of any dermatological or systemic disorder, which would have interfered with the results, at the discretion of the investigator.
3. Individuals who had completed a preliminary medical history mandated by Cantor Research Laboratories, Inc.
4. Individuals who had read, understood and signed an informed consent document as required by Reference 21 CFR Ch. 1 Part 50, Subpart B. Consent forms are kept on file and are available for examination on the premises of Cantor Research Laboratories, Inc., only.
5. Individuals who had abstained from the use of all moisturizing products for at least one week prior to treatment conditions.
6. Individuals with known dry skin.

Exclusion Criteria:

1. Individuals who were under doctor's care.
2. Individuals who were taking medication, which in the opinion of the investigator would have masked or interfered with the results.
3. Individuals with chronic skin allergies.
4. Females who were pregnant or lactating.

Ages: 35 Years to 57 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females only
Enrollment: 16 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Skin Hydration | Days 0, 7, 14 and 18
  Change in skin hydration (NovaMeter assessment)
Transepidermal water loss (TEWL) | Days 0, 14 and 18
  Change in transepidermal water loss (Vapometer assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Shyla Cantor, PhD, Study Director — Cantor Research Laboratory
Locations (1):
- Cantor Research Laboratory, Blauvelt, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be published in a scientific journal with raw data made available to researchers upon request.

REFERENCES:
- See also: Cantor Research Laboratory Website — http://www.cantorlabs.com/
- See also: Sytheon LTD Website — https://www.sytheonltd.com/